CLINICAL TRIAL: NCT06967077
Title: Exploring the Feasibility and Acceptability of Virtual Reality Exercise for Pain Management, Fear of Movement, Mobility, and Proprioception Deficit in Axial Spondyloarthritis Patients During Flares: Twics Design
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Alaa Jamil Kattan, Principal Investigator (PhD student), University of Bath
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 5485
Record Dates: First submitted 2025-03-26; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Axial Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Intervention Model Description: This study will employ the Trials within Cohort (TwiCs), which facilitates running an RCT by recruiting one control group for biomechanical and virtual reality assessments. From this group, eligible patients will be randomly selected to join the intervention arm, which involves a VR exercise intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention): Participants will undergo baseline assessments which includes:
  1. Spinal ROM and speed of movement, using a motion capture system (mocap)
  2. Questionnaires: BASFI, BASMI, BASDAI, TSK, PCS, VAS, and McGill Pain Questionnaire.
  3. JPE Testing: Proprioception will be assessed using VR system by targeting specific joint positions 10 times based on each participant's full ROM.
- Virtual reality group (Experimental): Participants will undergo baseline assessments which includes:
  1. Spinal ROM and speed of movement, using a motion capture system (mocap)
  2. Questionnaires: BASFI, BASMI, BASDAI, TSK, PCS, VAS, and McGill Pain Questionnaire.
  3. JPE Testing: Proprioception will be assessed using VR system by targeting specific joint positions 10 times based on each participant's full ROM.
  additionally they will be performing the VR tennis game for 10 minutes daily during flare stage.
  followed by feasibility assessment including usability and acceptability assessment of the VR intervention using both questionnaires and interviews during second and third sessions.
  Interventions: Other: Virtual reality head set.

INTERVENTIONS:
Other: Virtual reality head set. — Tennis game exercise using virtual reality head set
  Arms: Virtual reality group

SUMMARY:
Axial spondyloarthritis (axSpA) is an autoimmune disease that causes inflammatory arthritis of the spine, causing pain, stiffness, and mobility limitations. During flares, when symptoms worsen, people with axSpA often experience increased pain and difficulty moving, making daily activities more challenging. This study aims to explore whether virtual reality (VR) exercise can help manage pain, improve movement, and support rehabilitation for axSpA patients during flares.

Participants will use a VR system to perform gentle exercises designed to encourage movement and reduce discomfort. Their spinal mobility will be measured using motion capture technology, and their experiences with VR will be assessed through questionnaires and interviews.

This research will help determine whether VR can be a practical and beneficial tool for axSpA rehabilitation, potentially offering a new way to manage symptoms and improve quality of life. The findings will guide future studies on using VR in healthcare settings for people with chronic pain conditions.

DETAILED DESCRIPTION:
Axial spondyloarthritis (axSpA) is a chronic inflammatory disease affecting the spine and sacroiliac joints, causing pain, stiffness, and reduced mobility. Flares are periods of increased disease activity, which significantly impact patients' ability to move and perform daily tasks, often accompanied by heightened levels of pain and fear of movement, known as kinesiophobia., leading to long-term reductions in mobility and quality of life. Although physical activity is recognized as a valuable self-management tool, some axSpA patients report discomfort or joint injury during exercise, limiting their physical performance.

Additionally, proprioception is often impaired in inflammatory joint diseases, including axSpA. However, proprioception is poorly investigated in axSpA patients. There is a need to better understand mobility and proprioception during and after flares, as this could provide valuable insights for alleviating pain and enhancing functional mobility.

VR systems have shown promise in managing chronic pain and improving physical function through distraction and engaging virtual games. but its feasibility for axSpA patients remains understudied.

Aim:

Evaluate the feasibility of using VR exercises for axSpA patients during flare periods, for pain management, kinesiophobia, mobility improvement, and proprioception impairment.

Objectives:

1. To examine the impact of virtual reality (VR) training on reducing kinesiophobia, managing pain, and improving disease activity by analysing the correlation between range of motion (ROM) and velocity during VR training and the Tampa Scale of Kinesiophobia (TSK), Bath Ankylosing Spondylitis Functional Index (BASFI), Bath Ankylosing Spondylitis Metrology Index (BASMI), Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), Visual Analogue Scale (VAS), and McGill Pain Questionnaire.
2. To assess Proprioception with VR by joiny position error (JPE) test.
3. To evaluate the feasibility of using VR for axSpA rehabilitation by assessing usability and acceptability through interviews and questionnaires, including virtual reality sickness questionnaires and technology acceptance models (TAM).

This study will employ the Trials within Cohort (TwiCs), which facilitates running an RCT by recruiting one control group for biomechanical and virtual reality assessments. From this group, eligible patients will be randomly selected to join the intervention arm, which involves a VR exercise intervention.

All cohort participants will provide initial consent for the use of their observational data as controls. If selected for the intervention, additional consent will be obtained. Those allocated as controls will not need further consent and will continue with standard assessments.

Participants chosen for the intervention will receive an updated participant information sheet and will sign an additional consent form specific to the intervention.

All participants will attend four sessions: one at baseline, one during flare, one after flare, and one month post-flare.

Session 1 (Baseline Assessment): Participants will undergo baseline assessments which includes:

1. Spinal ROM and speed of movement, using a motion capture system (mocap)
2. Questionnaires: BASFI, BASMI, BASDAI, TSK, PCS, VAS, and McGill Pain Questionnaire.
3. JPE Testing: Proprioception will be assessed using VR system by targeting specific joint positions 10 times based on each participant's full ROM. participants will be randomly assigned to either the intervention group (VR) or the control group. Those in the intervention group will be informed of their eligibility and provided with an information sheet and consent form specific to the VR intervention. A demonstration of how to use the VR tennis game will be provided to ensure familiarity with the system.

Session 2 (During a Flare): All participants will complete the same assessments as in Session 1, with the intervention group additionally performing the VR tennis game followed by feasibility assessment including usability and acceptability assessment of the VR intervention using both questionnaires and interviews.

If a participant from the intervention group is unable to attend due to a severe flare, a VR headset will be delivered to their home along with a video tutorial to remind them of the previously demonstrated process. Both groups will complete BASDAI questionnaire daily using a link to Microsoft forms platform.

Session 3 (Post-Flare Assessment): Post-flare assessments will be conducted, including a repeat of baseline measures for both groups, and collection of participant feedback on the VR intervention through questionnaires and interviews for the intervention group..

Session 4 (One-Month Follow-up): A one-month follow-up assessment will be conducted repeating the assessment from first session for both groups.

Session 2 (During a Flare): All participants will complete the same assessments as in Session 1, with the intervention group additionally performing the VR tennis game. If a participant from the intervention group is unable to attend due to a severe flare, a VR headset will be delivered to their home along with a video tutorial to remind them of the previously demonstrated process. Both groups will complete BASDAI questionnaire daily using a link to Microsoft forms platform.

Session 3 (Post-Flare Assessment): Post-flare assessments will be conducted, including a repeat of baseline measures and the collection of participant feedback on VR usability.

Session 4 (One-Month Follow-up): A one-month follow-up assessment will be conducted to reassess mobility, pain, and proprioception outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of axial spondyloarthritis (axSpA).
2. Experiencing an active flare of axSpA within the last 6 months
3. Over 18 years of age.

Exclusion Criteria:

1. History of major spinal surgery.
2. Pregnancy.
3. Severe vestibular disorders, visual, balance, neurological, or cardiovascular conditions that may affect mobility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-10 (Estimated)

PRIMARY OUTCOMES:
1. Change in spinal mobility | between baseline and one month follow up
  Spinal mobility will be assessed using range of motion (ROM) measured via motion capture system.
Change in movement velocity | Baseline to one month follow up
  Movement velocity of spinal flexion, extension, and rotation will be measured using a motion capture system. Peak angular velocity (degrees/second) will be recorded during standardised movement tasks and compared between baseline and one-month follow-up.
  Unit of Measure: Degrees/second
Change in kinesiophobia | Baseline to one month follow up
  Kinesiophobia will be measured using the Tampa Scale of Kinesiophobia (TSK). The scale ranges from 17 to 68, with higher scores indicating greater fear of movement.
  Unit of Measure: TSK score (17-68; higher = worse)
Change in pain intensity | Baseline to one month follow up
  Pain intensity will be assessed using the Visual Analogue Scale (VAS). The scale ranges from 0 to 10, with higher scores indicating greater pain. Change from baseline to follow-up will be analysed.
  Unit of Measure: VAS score (0-10; higher = worse)
Changes in Pain severity and location | Baseline to one month follow up
  Pain severity and location will be assessed using the McGill Pain Questionnaire Short Form (MPQ-SF). The scale ranges from 0 to 78, with higher scores indicating greater pain severity.
  Unit of Measure: MPQ-SF score (0-78; higher = worse)
proprioception impairment | from baseline to one month follow up.
  Changes in JPE scores between flare and non-flare stages to determine proprioception impairments
  Joint Position Error (JPE) will be measured using a spine movement reposition task by asking participants to duplicate angle of movement (for example 45 degree of spine flexion) to assess spine proprioception. Higher JPE scores reflect greater proprioceptive impairment.
  Unit of Measure: Degrees of deviation from target position Scale Range: 0-180 degrees (theoretically depends on direction of movement); lower scores indicate better proprioception
Change in spinal flexibility | Baseline to one month follow up
  Spinal flexibility will be measured using the Bath Ankylosing Spondylitis Metrology Index (BASMI). The scale ranges from 0 to 10, with higher scores indicating worse spinal mobility.
  Unit of Measure: BASMI score (0-10; higher = worse)
Change in Disease Activity | Baseline to one month follow up
  Improvement in disease activity assessed using the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Change in Functional Limitation | from baseline to one month follow up.
  Improvement in functional limitation as assessed by the Bath Ankylosing Spondylitis Functional Index (BASFI) and its correlation with objective movement parameters.
  BASFI (0-10 scale): Higher scores indicate worse functional limitation.
Usability of VR rehabilitation | from baseline to one month follow up.
  Usability will be assessed using the System Usability Scale (SUS).
  SUS: A 10-item scale with scores ranging from 0 to 100. Higher scores indicate better usability.
  Unit of Measure: SUS score (0-100)
Motion Sickness Symptoms During VR Use | Baseline to one month follow up
  motion sickness, will be assessed using the Virtual Reality Sickness Questionnaire (VRSQ).
  VRSQ: Includes multiple subscales measuring symptoms such as oculomotor strain and disorientation.
  Higher scores indicate greater motion sickness symptoms.
  Unit of Measure: VRSQ subscale scores
Acceptability of VR Rehabilitation | Baseline to one month follow up
  Acceptability will be assessed through semi-structured interviews exploring participants' experiences, perceived benefits, barriers to use, and overall views on the intervention.
  Unit of Measure: Qualitative themes derived from participant interviews

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including movement analysis, pain scores, and patient-reported outcomes, will be shared exclusively with my PhD supervisors for internal review and guidance. No public access or external data requests will be permitted. Personal identifiers will be removed to maintain confidentiality
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be made available to supervisors during the study period and up to one year after completion for internal review and analysis
Access Criteria: Access is restricted to my PhD supervisors for internal study review. No external sharing will be permitted. The data will be handled in accordance with institutional and ethical guidelines

REFERENCES:
- [Background] Hoffman HG, Patterson DR, Carrougher GJ, Sharar SR. Effectiveness of virtual reality-based pain control with multiple treatments. Clin J Pain. 2001 Sep;17(3):229-35. doi: 10.1097/00002508-200109000-00007. PMID 11587113
- [Background] Seerden SFL, Dankaerts W, Swinnen TW, Westhovens R, De Vlam K, Vanwanseele B. Axial Spondyloarthritis is associated with changes in lumbosacral loading during daily activities. Clin Biomech (Bristol). 2021 May;85:105347. doi: 10.1016/j.clinbiomech.2021.105347. Epub 2021 Apr 3. PMID 33905963
- [Background] Seerden SFL, Dankaerts W, Swinnen TW, Westhovens R, De Vlam K, Vanwanseele B. Differences in multi-segmental spine kinematics between patients with different stages of axial spondyloarthritis and healthy controls. Musculoskelet Sci Pract. 2021 Jun;53:102368. doi: 10.1016/j.msksp.2021.102368. Epub 2021 Mar 19. PMID 33780698
- [Background] Mouatt, B., Smith, A.E., Mellow, M.L., Parfitt, G., Smith, R.T. and Stanton, T.R., 2020. The use of virtual reality to influence motivation, affect, enjoyment, and engagement during exercise: A scoping review. Frontiers in Virtual Reality, 1, p. 564664.
- [Background] Ozen T, Tonga E, Polat MG, Bayraktar D, Akar S. Cervical proprioception accuracy is impaired in patients with axial spondyloarthritis. Musculoskelet Sci Pract. 2021 Feb;51:102304. doi: 10.1016/j.msksp.2020.102304. Epub 2020 Nov 16. PMID 33227676
- [Background] Barnett R, Ng S, Sengupta R. Understanding flare in axial spondyloarthritis: novel insights from daily self-reported flare experience. Rheumatol Adv Pract. 2021 Nov 15;5(3):rkab082. doi: 10.1093/rap/rkab082. eCollection 2021. PMID 34926981
- [Background] Aouad K, Gossec L. Defining and managing flares in axial spondyloarthritis. Curr Opin Rheumatol. 2022 Jul 1;34(4):195-202. doi: 10.1097/BOR.0000000000000883. Epub 2022 Jun 9. PMID 35699318